CLINICAL TRIAL: NCT00698269
Title: Efficacy and Safety Study in Subjects Using Levemir® (Insulin Detemir), NovoMix®30 (Biphasic Insulin Aspart 30) and/or NovoRapid® (Insulin Aspart) for the Treatment of Type 1 or Type 2 Diabetes Mellitus
Brief Title: An Observational Study of Efficacy and Safety of Modern Insulin in Diabetes Patients Switched From Anti-diabetic Treatment
Status: Completed | Type: Observational
Sponsor: Novo Nordisk A/S (Industry)
Responsible Party: Sponsor
Other Study IDs: INS-3532
Record Dates: First submitted 2008-06-13; First posted 2008-06-17 (Estimated); Last update posted 2016-10-28 (Estimated); Status verified 2016-10

CONDITIONS: Diabetes; Diabetes Mellitus, Type 1; Diabetes Mellitus, Type 2
MeSH Terms: conditions — Diabetes Mellitus; Diabetes Mellitus, Type 1; Diabetes Mellitus, Type 2 | interventions — Insulin Detemir; insulin aspart, insulin aspart protamine drug combination 30:70; Insulin Aspart

STUDY DESIGN:
Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (3):
- A
  Interventions: Drug: insulin detemir
- B
  Interventions: Drug: biphasic insulin aspart 30
- C
  Interventions: Drug: insulin aspart

INTERVENTIONS:
Drug: insulin detemir — Start dose and frequency to be prescribed by the physician as a result of the normal clinical evaluation
  Other Names: Levemir®
  Groups: A
Drug: biphasic insulin aspart 30 — Start dose and frequency to be prescribed by the physician as a result of the normal clinical evaluation
  Groups: B
Drug: insulin aspart — Start dose and frequency to be prescribed by the physician as a result of the normal clinical evaluation
  Groups: C

SUMMARY:
This study is conducted in Asia. The aim of this observational study is to evaluate the safety and efficacy of modern insulins after switch from any other anti-diabetic treatment under normal clinical conditions in the Gulf countries.

ELIGIBILITY:
Inclusion Criteria:

* Type 1 or type 2 diabetes
* Treatment with any diabetes treatment other than NovoMix® 30, Levemir® and/or NovoRapid®
* Selection will be at the discretion of the individual physician

Exclusion Criteria:

* Current treatment with Levemir®, NovoMix® 30 and/or NovoRapid®
* Previous enrolled in this study
* Hypersensitivity to Levemir®, NovoMix® 30 and/or NovoRapid® or to any of the excipients
* Women who are pregnant, breast feeding or have the intention of becoming pregnant within next 6 months

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: A non-randomized sample of Type 1 or Type 2 diabetics
Sampling Method: Probability Sample
Enrollment: 5926 (Actual)
Dates: Start 2008-02; Primary Completion 2009-08 (Actual); Study Completion 2009-08 (Actual)

PRIMARY OUTCOMES:
Incidence of major hypoglycaemic events reported | during 24 weeks of treatment
Change in HbA1c | during 24 weeks of treatment

SECONDARY OUTCOMES:
Percentage of subjects achieving HbA1c below 7.0% | at 12 & 24 weeks
Change in FPG | at 12 & 24 weeks
Change in PPG | at 12 & 24 weeks
Body weight | at 12 & 24 weeks
Change in number of hypoglycaemic events in the last 4 weeks before routine visits | at 12 & 24 weeks
Change in number of nocturnal Hypoglycaemic events in the last 4 weeks before routine visits | at 12 & 24 weeks
Number of adverse drug reactions (ADR) | at 12 & 24 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Global Clinical Registry (GCR, 1452), Study Director — Novo Nordisk A/S
Locations (1):
- Novo Nordisk Investigational Site, Riyadh, Saudi Arabia

REFERENCES:
- See also: Clinical Trials at Novo Nordisk — http://novonordisk-trials.com